CLINICAL TRIAL: NCT03795883
Title: The Thrombotic Potential (Thrombin Generation) of Left Atrium and Other Heart Chambers in Atrial Fibrillation Patients Compared to Patients Without Atrial Fibrillation.
Brief Title: The Thrombotic Potential of Heart Chambers in the Presence or Absence of Atrial Fibrillation.
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Adi Elias MD, Resident Physician at Cardiology Department, Principal Investigator, Rambam Health Care Campus
Other Study IDs: RMB CTIL-0216-18
Record Dates: First submitted 2018-12-30; First posted 2019-01-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation; Thrombosis Cardiac; Left Atrial Thrombosis
Keywords: Thrombin generation; Calibrated automated thrombogram; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ten cc of blood will be collected from each heart chamber (Left atrium, Left atrial appendage, Right atrium, Right ventricle) and peripheral vein
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with atrial fibrillation: Patients with atrial fibrillation admitted for standard pulmonary vein ablation.
- Participants without atrial fibrillation: Patients without atrial fibrillation admitted for standard left sided supra ventricular tachycardia ablation or patients admitted to mitral clip procedure.

SUMMARY:
The investigators aim to test the thrombotic potential of various heart chambers including left atrium, left atrial appendage, right atrium and peripheral veins. Blood samples will be taken from the different chambers in 50 patients admitted for standard pulmonary vein ablation and compared to patients without atrial fibrillation admitted for left sided supra ventricular tachycardia or mitral clip. Thrombin generation parameters will be assessed by the calibrated automated thrombogram.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common arrhythmia, there is a strong correlation between atrial fibrillation and embolic stroke. In order to lower the risk for embolic stroke anticoagulation is recommended for patients with CHADS-VASC score equal or above 2. The mechanism for thrombus formation in the left atrium is thought to be caused by various factors 1. blood stasis due to the loss of atrial kick 2. endothelial dysfunction 3. blood hemostatic alteration leading to procoagulant state.

Previous studies demonstrated increased thrombin generation in the left atrium in patients with atrial fibrillation, when compared to other heart chambers and when compared to control group in patients with structurally normal heart.

In recent years calibrated automated thrombogram (CAT) is considered a good indicator for total thrombotic activity in hypercoagulable states.

In the current study the investigators aim to test the thrombotic potential of various heart chambers including left atrium, left atrial appendage, right atrium and peripheral veins. Blood samples will be taken from the different chambers in 50 patients admitted for standard pulmonary vein ablation without changing the course of the procedure. Thrombin generation parameters will be assessed by the calibrated automated thrombogram. A control group composed of 50 patients admitted for standard left sided supra ventricular tachycardia ablation or patients admitted to mitral clip procedure without the presence of atrial fibrillation.

In addition demographic data,CHADS-VASC score, atrial fibrillation burden, echocardiographic and cardiac CT parameters will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Pulmonary vein ablation, SVT ablation or mitral clip.
* Informed consent

Exclusion Criteria:

* Left atrial thrombus
* Pregnancy
* Active malignancy
* Thrombophilia
* Anticoagulants 24 hours before procedure
* Active infectious disease
* Chronic kidney disease (eGFR<30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group:Participants with atrial fibrillation admitted to pulmonary vein ablation Control group: Participant without atrial fibrillation admitted to left sided SVT ablation or Mitral clip.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
ETP of various heart chambers measured by the calibrated automated thrombogram (CAT) | 1 Day
  ETP (endogenous thrombotic potential) nM*min
Peak height of various heart chambers measured by the calibrated automated thrombogram (CAT) | 1 Day
  Peak height nM
Lag time of various heart chambers measured by the calibrated automated thrombogram (CAT) | 1 Day
  Lag time in minutes
Time to peak of various heart chambers measured by the calibrated automated thrombogram (CAT) | 1 Day
  Time to peak in minutes

SECONDARY OUTCOMES:
The 1 year incidence of thromboembolic events | 1 Year
The number of participants with spontaneous echocardiographic contrast demonstrated in trans-esophageal echocardiogram (TEE) | 1 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elias A, Khoury Y, Shehadeh F, Ron G, Boulos M, Nashashibi J, Zukermann R, Elias M, Gepstein L, Suleiman M. Elevated thrombin generation levels in the left atrial appendage in patients with atrial fibrillation. Res Pract Thromb Haemost. 2023 Mar 15;7(2):100127. doi: 10.1016/j.rpth.2023.100127. eCollection 2023 Feb. PMID 37063762